CLINICAL TRIAL: NCT03619304
Title: Assessment of Anti-cancerous Effect of Green, Roasted and Decaffeinated Coffee on Oral Squamous Cell Carcinoma Cell Line
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Emad El- Din Mohammed, Teaching assistant oral pathology department, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-7-02
Record Dates: First submitted 2018-07-06; First posted 2018-08-07 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: coffee, oral squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Coffee

STUDY DESIGN:
Intervention Model Description: oral squamous cell carcinoma cell lines
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- no coffee (Experimental): oral squamous cell carcinoma cell line without intervention
  Interventions: Dietary Supplement: coffee
- green coffee (Active Comparator): oral squamous cell carcinoma cell line with application of green coffee
  Interventions: Dietary Supplement: coffee
- roasted coffee (Active Comparator): oral squamous cell carcinoma cell line with application of roasted coffee
  Interventions: Dietary Supplement: coffee
- decaffeinated coffee (Active Comparator): oral squamous cell carcinoma cell line with application of decaffeinated coffee
  Interventions: Dietary Supplement: coffee

INTERVENTIONS:
Dietary Supplement: coffee — coffee beverage

SUMMARY:
Oral cancer is the sixth most common cancer worldwide. Over 90% of all identified oral cavity cancers are invasive oral squamous cell carcinomas (OSCCs). Primary treatments of OSCC are surgery, radiation therapy, and chemotherapy. However, anticancer therapies (drugs, irradiation) have undesirable side effects as they may induce mutations or irreversible DNA damage killing healthy cells.

One of the most frequently used alternative therapies is herbal medicine that act as anti-ROS agents preventing DNA damage has been used alongside conventional treatment regimens. One of the agents that receives particular strong interest is coffee. Coffee is considered as a major source of dietary antioxidants; some are present in the green bean, whereas others are generated during roasting. Coffee roasting, the process of the heating of green coffee beans transforming them into black coffee beans, transforms the chemical and biological properties of coffee beans.

Regarding oral cancer, some studies reported an association of high coffee consumption to an augmented risk of oral cancer while others showed a clear inverse association with the risk of oral cancer. Recently, there have been reports of a protective effect of coffee consumption on oral cancer from two recent meta-analysis. To our knowledge, only two studies were done to assess the effect of coffee ingredients (cafestol and kahweol) on oral squamous cell carcinoma cell lines.

Due to these controversial findings concerning the effect of roasted coffee and absence of data on unprocessed (green coffee), our study aims to investigate the effect of different coffee beverage as regard apoptosis and proliferation carried out in OSCC cell lines.

DETAILED DESCRIPTION:
Oral cancer is the sixth most common cancer in males and the twelfth most common in females. Approximately, 94% of all oral malignancies are squamous cell carcinoma. Over the past few decades, researchers have explored alternate therapies and remedies to prevent its progression but have yielded to low success rates. Targeted therapy of oral cancer is promising following identification of anticancer biomolecules. Naturally available extracts have been desired after in this regard as an adjunctive therapeutic modality.

Current research in the head and neck cancer mainly focuses to understand the molecular mechanisms of oral cancer development and progression to target the biomarkers and facilitate the development of new treatment strategies. Studies with cell lines can serve as an initial screen for agents that might regulate drug resistance and to establish whether the differences exist in the different drug-resistant sublines.

Phytochemicals and extracts derived from medicinal plants have been noted as promising cancer-preventive agents against several cancers because of their low toxicity and the accumulating data supporting their beneficial health effects. Coffee, after water, is the leading beverage in the world which highlights the importance of knowledge of its possible influence on human health. Coffee beverages contain a variety of antioxidant and antimutagen agents including phenolic derivatives such as chlorogenic acid and polyphenol caffeic acid and diterpenes such as cafestol and kahweol. Some studies have suggested that these constituents could provide some genotoxicity protection thus classifying coffee as anti-cancer agent. However, future work in the mechanism is needed because coffee has many components, and effects may depend on multiple factors such as the type of coffee bean, caffeinated compared with decaffeinated coffee, roasting, and brewing methods.

Several studies have tried to analyze the contribution of coffee consumption on the risk of different cancer types. The effect of coffee on cancer risk is controversial because both inhibiting and promoting effects have been suggested. The antioxidative effect of chlorogenic acid and the inhibitory effect of DNA methylation are considered to contribute to coffee's protective effect.

A protective effect of coffee has been observed in humans for a variety of cancers. The most recent studies have reported that coffee is inversely associated with oral cancer/pharyngeal cancer, basal cell carcinoma and endometrial cancer type I. Coffee drinking has been also inversely related to colorectal cancer and liver cancer. However, the caffeine in coffee is known to modify the apoptotic response and disturb cell checkpoint integrity.

The type of coffee has a significant impact on their antioxidant potential. Thermal treatment of coffee beans (roasting process) also affects the level of antioxidant potential. Roasting process transforms the chemical and biological properties of coffee beans and increases its antioxidant activity. Roasted coffee beans exhibited higher antioxidant capacity than green coffee beans, and intensified coffee roasting resulted in a decrease of its antioxidant potential.

To our knowledge, only one study which reported the effect of different types of coffee beverage (caffeinated, decaffeinated and coffee) on oral cancer risk. Besides, the evidence of the effect of green coffee and decaffeinated coffee on OSCC was very scarce. The exact biological mechanism of potentially healthy role of coffee in head and neck cancer is still not available.

ELIGIBILITY:
Inclusion Criteria:

* human cell lines
* only oral squamous cell carcinoma cell line
* green coffee extract
* roasted coffee extract
* decaffeinated coffee extract

Exclusion Criteria:

- mixed tumors animal cell lines

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-07-17 (Estimated)

PRIMARY OUTCOMES:
Apoptotic cell death | 3 months
  Apoptosis

CONTACTS AND LOCATIONS:
Overall Officials: Manar M Abd el wanis, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03619304/Prot_000.pdf